CLINICAL TRIAL: NCT06131099
Title: Effects of Dohsa Hou Exercises on Functional Mobility in Children With Down Syndrome
Brief Title: Effects of Dohsa Hou Exercises on Functional Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0762
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
Keywords: Dohsa hou exercise; Down syndrome; Psychomotor therapy
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Its a randomized control trail, used to compare the effects of Dohsa hou exercises on functional mobility in children with Down syndrome. Subjects with Down syndrome meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): In this group patient will be treated with standard treatment protocol. This group will receive therapy session for 1 hour, three sessions in a week and for 6 weeks, total sessions will be 18. Group A will receive soft tissue massage therapy for 5 mins and the task specific training interventions include bicycle training for 10 mins. After that aerobic exercises includes and finally some of progressive resistive exercises will involve in it.
  Interventions: Other: Standard treatment protocal
- Group B (Active Comparator): In this group patient will be treated with Dohsa hou exercises. This group will receive therapy session for 1 hour, three sessions in a week and for 6 weeks, total sessions will be 18. Group B will receive Dohsa hou exercises, session will be included three activity parts: (a) 10 minutes of instruction and preparation, (b) 45 minutes of skill instruction and practice, and (c) 5 minutes in a closing activity.
  Interventions: Other: Dohsa hou exercises

INTERVENTIONS:
Other: Dohsa hou exercises — Dohsa hou is a type of psychomotor therapy that helps improve psychological problems by using bodily movements, sensation and relaxation experience.
  Arms: Group B
Other: Standard treatment protocal — Standard treatment including soft tissue massage therapy, task specific training interventions, bicycle training and aerobic exercises.
  Arms: Group A

SUMMARY:
Trisomy 21 is a condition where there's an extra chromosome 21, which leads to a set of clinical signs called Down syndrome. Down syndrome is one of the most complicated genetic conditions that can occur post-term and is the most commonly survivable form of aneuploidy of the autosomal chromosomes.

Dohsa hou is a type of psychomotor therapy that helps improve psychological problems by using bodily movements, sensation and relaxation experience. It was first developed under the name psycho-rehabilitation to help children with cerebral palsy improve their movements and posture. By using Dohsa hou movement's issues were effectively addressed in children with cerebral palsy, despite their physical limitations being caused by physiological disorders. There are two kind of treatments of Dohsa hou exercises that are relaxation therapy to decrease the stress level in body and other one is to align the body to correct the posture and movements of the body.

DETAILED DESCRIPTION:
This study will be a randomized control trial, used to compare the effects of Dohsa hou exercises on functional mobility in children with Down syndrome. Subjects with Down syndrome meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling techniques. Assessment will be done by using Test of trunk impairment scale and Time Up and Go Test. Subjects in one group will be treated with Dohsa hou therapy and in other group standard treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Down syndrome
2. Age group of 6 to 12 years old
3. Male and female (both genders)
4. Body mass index (BMI) within normal range <95%
5. Absence of any psychiatric and physical illness at the time of participation.

Exclusion Criteria:

1. Uncontrolled seizures
2. Any kind of autoimmune diseases
3. Registered visually impaired or hearing issues
4. Severe atlanto axial instability
5. Congenital heart defects (CHD)
6. Unable or unwilling to understand the commands

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Trunk impairment scale | 6 weeks
  The trunk impairment scale will be used for this study to identify the balance and coordination in sitting and standing state. The assessment tool uses a 2 to 4 point ranking system for each item. The highest possible scores for the static and dynamic sitting balance and coordination scales are 7, 10 and 6 points. The TSI score can range from 0 to 23, with a score of 0 indicating minimal performance and a perfect score of 23.
Time up and go | 6 weeks
  Time up and go test will be used to assess the balance and stability of a children with different abilities. It involves timing how long it takes for a child to stand up from a chair, walk a short distance, turn around, walk back, and sit down while turning 180 degree.
  Interpretation: < 10 seconds = normal, < 20 seconds = good mobility, can go out alone, mobile without a gait aid. < 30 seconds = problems, cannot go outside alone, requires a gait aid. A score of more than or equal to fourteen seconds has been shown to indicate high risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asif Javed, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fujino H, Moritsugu A. Dohsa-hou for unexplained regression in Down syndrome in a 19-year-old man: A case report. Clin Case Rep. 2022 May 15;10(5):e05827. doi: 10.1002/ccr3.5827. eCollection 2022 May. PMID 35600012